CLINICAL TRIAL: NCT06604546
Title: Pharmacodynamic Clinical Trail of Recombinant Human Hyaluronidase Assisted Subcutaneous Infusion in Healthy Volunteers
Brief Title: Hyaluronidase Assisted Subcutaneous Infusion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Bao Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHBJ-KJ017-001
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Healthy
MeSH Terms: interventions — Hyaluronoglucosaminidase; Ringer's Lactate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hyaluronidase group (Experimental)
  Interventions: Drug: hyaluronidase
- Placebo self control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hyaluronidase — 150 IU group D1:150 IU hyaluronidase+500 ml Lactated Ringer's (LR)(Subject's left or right leg)； D2:150 IU hyaluronidase+250 ml Lactated Ringe's (LR)(Subject's left or right arm)； D3:150 IU hyaluronidase+500 ml Normal Saline (NS)(subject's left or right leg)； D4:150 IU hyaluronidase+1000 ml Lactated Ringer's (LR)(Subject's back)； 385 IU group D1:385 IU hyaluronidase+250 ml Lactated Ringer's (LR)(Subject's left or right arm)； 1500 IU group D1:1500 IU hyaluronidase+250 ml Lactated Ringer's (LR)(Subject's left or right arm).
  Other Names: Lactated Ringer's (LR); Normal Saline (NS)
  Arms: hyaluronidase group
Drug: Placebo — 150 IU group D1:Placebo+500 ml Lactated Ringer's (LR)(Subject's left or right leg)； D2:Placeboe+250 ml Lactated Ringer's (LR)(Subject's left or right arm)； D3:Placebo+500 ml Normal Saline (NS)(Subject's left or right leg)； 385 IU group D1:Placebo+250 ml Lactated Ringer's (LR)(Subject's left or right arm)； 1500 IU group D1:Placebo+250 ml Lactated Ringe's (LR)(Subject's left or right arm).
  Other Names: Lactated Ringer's; Normal Saline
  Arms: Placebo self control group

SUMMARY:
A randomised, double-blind, self controlled study to evaluate the pharmacodynamics and safety of recombinant human hyaluronidase assisted subcutaneous infusion in healthy subjects.

Recombinant human hyaluronidase or placebo was injected subcutaneously at the prescribed site on the day of administration. The prescribed fluid was then infused subcutaneously.

Subjects in the 150 IU group received a subcutaneous infusion of 500 mL Ringer's lactated sodium into the lateral thighs bilaterally on D1, 250 mL Ringer's lactated sodium into the upper arms bilaterally on D2, 500 mL sodium chloride injection into the lateral thighs bilaterally on D3, and 1,000 mL Ringer's lactated sodium into the back on D4, as scheduled.

Subjects in the 385 IU group received a 250 mL subcutaneous infusion of Ringer's lactated sodium into the bilateral upper arms on D1 as scheduled.

Subjects in the 1500 IU group received a 250 mL subcutaneous infusion of Ringer's lactated sodium into the bilateral upper arms on D1 as scheduled.

DETAILED DESCRIPTION:
Hyaluronic acid (HA) is an acidic mucopolysaccharide widely found in connective tissues such as the intercellular matrix of human tissues, the vitreous humour of the eye and the synovial fluid of the joints, and is a component of the tissue matrix that acts to restrict the diffusion of water and other extracellular substances. Its gel-like nature makes it a barrier to subcutaneous fluid diffusion and is an important limitation to subcutaneous infusion. It has also been reported in the literature that lymph nodes, liver and skin are the major metabolic sites of HA, with a metabolic half-life in the skin of approximately 15-20 h. This means that the structure of HA destroyed by enzymatic cleavage can be autonomously rebuilt within 24-48 h. The rapid metabolism characteristics of HA make it an ideal target for action. Hyaluronidase is an endoglycosidase capable of degrading and oligomerising HA. HAase hydrolyses the β-1,4 glycosidic linkage in the HA chain to yield small molecules of HA or oligosaccharides, thereby increasing tissue permeability and improving the permeability of tissues to fluids. HAase has been used in the medical field for many years as a drug diffusing agent, which can promote the diffusion of locally stored drugs, exudate or blood, accelerate the absorption of drugs, reduce local tissue tension and pain, and facilitate the absorption and drainage of oedema and inflammatory exudate. Clinically, HAase is used clinically as an adjunct to subcutaneous infusion.

ELIGIBILITY:
Inclusion criteria:

1. Must be willing to participate in this study and sign a written informed consent form.
2. Male or female, 18 to 60 years of age.
3. Male subjects weighing at least 50 kg, female subjects weighing at least 45 kg. Body mass index in the range of 18-28 kg/m2 (including threshold values).

Exclusion criteria:

1. Positive for HBsAg, HCV antibody, HIV antibody and syphilis antibody at screening.
2. Definite hypersensitivity to recombinant human hyaluronidase for injection or any of the components of its preparation. Severe allergic reaction (e.g. angioedema) to any medication. Special dietary requirements or inability to follow the standard diet required by the clinical trial site.
3. Prescription medicines taken within 14 days or 5 half-lives prior to dosing, or over-the-counter medicines (including proprietary Chinese medicines and herbal remedies) taken within 7 days or 5 half-lives prior to dosing. Regular vitamin supplementation was excluded, but special cases of medication that, in the opinion of the investigator, did not interfere with the evaluation of the study could be included.
4. Blood donation or blood loss of 400 mL or more in the 3 months prior to screening.
5. Heavy smoking (25 or more cigarettes per day).
6. Alcohol abuse or a positive breath test result for alcohol.
7. Positive urine drug screen (including morphine, methamphetamine, ketamine).
8. Received another investigational drug (or investigational device) within 28 days or at least 5 half-lives prior to screening, whichever is longer.
9. The subject or partner is planning to have a child or is unwilling to use effective contraception during the trial or for 6 months after the end of the trial.
10. Nursing or pregnant women.
11. Inflammation, tattoos, skin lesions, and scarring on both limbs may interfere with observation and assessment.
12. Extremities oedema and limb pathology that may affect test results (e.g. cellulitis, lymphatic disorders or history of surgery, history of mastectomy, history of pre-existing pain syndrome or axillary lymph node dissection).
13. Sensorimotor and voluntary movement disorders.
14. Circumstances such as the investigator's opinion that participation in the trial is inappropriate or that the subject is unable to participate in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Subcutaneous infusion rate. | Within 4 hours after starting subcutaneous infusion.
  Subcutaneous infusion Rate: defined as Infusion Rate = (Base Infusion Bag Weighing Weight - Final Infusion Bag Weighing Weight) x (1 mL/g)/(Infusion Completion Time - Infusion Start Time).

SECONDARY OUTCOMES:
Immunogenicity | day 21
  antidrug antibodies (ADA) level
Measurement value of limb circumference | day 4
  Limb circumference measurements: Limb circumference measurements were used to assess the pharmacodynamic and safety profile of subcutaneous infusions in healthy volunteers. Limb circumference was measured at the time of each subcutaneous infusion in the upper arm or thigh and at the end of the infusion until the limb circumference returned to baseline (±2 cm).
Adverse events | day 7
  The Investigator will carefully monitor each subject throughout the study for any adverse events (coded to preferred term and system organ class using the Medical Dictionary for Regulatory Activities [MedDRA]). Adverse events assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Municipal Hospital, Suzhou, Jiangsu, China